CLINICAL TRIAL: NCT05041166
Title: Optimized In-Human [13C]Pyruvate MRI For Assessment Of Physiologic Reference Data In Different Organs
Brief Title: A Study of [13C]Pyruvate as an Imaging Agent for Magnetic Resonance Imaging in Healthy Volunteers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-309
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: MRI; Hyperpolarized (HP) [13C] pyruvate; 21-309
MeSH Terms: interventions — Pyruvic Acid

STUDY DESIGN:
Intervention Model Description: This in-human study of HP [13C]pyruvate MRI at MSKCC will be an open-label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Protocol optimization cohort (Experimental): Following the [13C]pyruvate injection, dynamic imaging and 3D volumetric imaging of volunteers in the first cohort (HP MRI protocol optimization, Aim 1) will be performed on the 3-T MRI scanner, using different [13C] RF excitation/detection coils.
  Interventions: Drug: Hyperpolarized [13C] Pyruvate
- Tissue reference cohort (Experimental): The optimal setup will then be used for HP MRI of the second cohort.
  Interventions: Drug: Hyperpolarized [13C] Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized [13C] Pyruvate — Will be injected at a dosage of 0.43 ± 0.05 mL/kg body weight

SUMMARY:
The purpose of the study is to learn about the use of [13C]pyruvate as an imaging agent for MRI scans. In past studies, researchers have seen that [13C]pyruvate can improve imaging with MRI scans. However, they would like to know more about how the imaging agent is distributed in healthy organs and tissues. This study will provide additional information about the use of [13C]pyruvate as an imaging agent for MRI scans, and it will show us how the substance is metabolized (changed into energy) in the organs and tissues of healthy volunteers. For (n=5) volunteers undergoing brain imaging we will compare the standard injection at 5mL/second with a slower infusion (0.1-1mL/second) to achieve a 60 second infusion time, to approach quasi steady-state metabolism and improve SNR.

ELIGIBILITY:
Inclusion Criteria:

Fifty healthy volunteers will be included.

* Age between 18-80
* Negative serum or urine pregnancy test for female volunteers of childbearing age and potential (as defined by MSKCC Standards & Guidelines), from assays obtained <2 weeks prior to study enrollment. Urine pregnancy tests are only valid for the day of test.

Exclusion Criteria:

* Breast-feeding
* History of metabolic (e.g. diabetes) and renal functional disorders.
* Refusal or inability to tolerate the scanning procedure (e.g., due to claustrophobia)
* Acute major illness (e.g., unstable cardiovascular condition, systemic malignant diseases, etc.).
* Standard MRI safety screening will be applied (MRI screening questionnaire); volunteers with MR unsafe devices, or conditional devices where research mode is not allowed, will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratios | 1 day
  will be used to assess image quality, and to compare the different technical setups. The setup providing the highest SNR will be considered optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Vesselin Miloushev, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm